CLINICAL TRIAL: NCT04658264
Title: Nutrient Profiling and Bio-efficacy of an Economic and Palatable Composite Flour for Type-2 Diabetes and Associated Metabolic Abnormalities in Open Label Randomized Control Clinical Trial
Brief Title: Nutrient Profiling and Bio-efficacy of Wheat-Barley Composite Flour in Type-2 Diabetes a in Randomized Control Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 039/IRC/BMR
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Barley/Wheat Composite Flour in Type-2 Diabetes
Keywords: Barley in Diabetes, Composite flour in Diabetes, Beta Glucan in Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): The Treatment group shall receive 2 Kg of the composite flour every week, sufficient for 21 chapattis, and shall eat chapattis made from this flour instead of their usual wheat flour chapattis. The participants shall continue to receive the usual treatment suggested by their physician along with any changes that the physician deems necessary during the 3 month period of this study.
  Interventions: Dietary Supplement: Wheat-Barley Composite flour
- Control Group (No Intervention): This group shall receive only the usual treatment suggested by their physician along with any changes that the physician deems necessary during the 3 month period of this study. They will continue to eat their usual diet as before their enrollment. They shall however receive usual counseling on lifestyle modifications including diet

INTERVENTIONS:
Dietary Supplement: Wheat-Barley Composite flour — A combination of wheat and barley flour with 0.5% food grade xanthan gum as replacement for lost gluten, tested for sensory properties, nutrient profile, and rheology
  Arms: Treatment Arm

SUMMARY:
Diabetes is a chronic disorder of metabolism characterized by hyperglycemia, defect in Insulin secretion, defection in Insulin action or both, which has a high potential for serious complications with high mortality and morbidity, if poorly treated. Outcome improves with better control.

It is a very common disorder with current global prevalence of 425 million and the latest diabetes survey of Pakistan in 2017-18 shows a prevalence of 26 % in adults.

Lifestyle intervention especially nutritional modification was the earliest intervention tried and still relevant. Strict Diet plans are difficult to follow; hence a functional Food based intervention is more likely to be acceptable. Various functional foods have been tried in diabetes but beta glucan , a soluble fiber found in barley has been widely tested and found to be effective not only in controlling glycemia, but also in improvement of dyslipidemia, blood pressure and weight.

This study has been planned with the objectives of formulating a composite flour based on wheat and barley, which is palatable, economical and can be used instead of wheat flour in the routine diet of people with diabetes.Xanthan Gum shall be added to compensate for the gluten loss. Various ratios of the flour shall be tested for sensory qualities, rheology, and glycemic index, and beta glucan content, and an acceptable flour with best attributes shall be further evaluated through proximate analysis and finally tested in a randomized in an open label randomized controlled clinical trial in real patients at Akhuwat Medical Center which is a charity facility.The sample size for a power of 90 has been calculated to be 31 and adding for dropouts , rounded up to 35 for each group. 70 Adult non pregnant Type 2 Diabetics above the age of 25, with no serious comorbidity shall be recruited and randomized through computer generated random number table. One group shall receive the 2 kg of composite flour every week for 3 months in addition to usual treatment while the con troll group shall receive only the usual treatment.

BMI, HbA1C, Creatinine, fasting lipid profile and ALT shall be measured at the start and end of the study, while ,Fasting and post meal sugars, BP, appetite, satiety, and compliance shall be measured every week. The data shall be processed in SPSS 23 This study is expected to show a significant improvement in glycemic control with a possible benefit in BP, weigh and lipid profile as well

DETAILED DESCRIPTION:
Background: Diabetes is a chronic disorder of metabolism characterized by hyperglycemia, defect in Insulin secretion, defect in Insulin action or both, which has a high potential for serious complications with high mortality and morbidity, if poorly treated. Outcome improves with better control. It is a very common disorder with current global prevalence of 425 million and the latest diabetes survey of Pakistan in 2017-18 shows a prevalence of 26 % in adults. Lifestyle intervention especially nutritional modification was the earliest intervention tried and still relevant. Strict Diet plans are difficult to follow; hence a functional food based intervention is more likely to be acceptable. Various functional foods have been tried in diabetes but beta glucan, a soluble fiber found in barley has been widely tested and found to be effective not only in controlling glycemia, but also in improvement of dyslipidemia, blood pressure and weight.

Hypothesis: Wheat-barley composite flour replaced with wheat in the diet of diabetics will improve their glycemic control.

Methodology: The study shall be conducted in two phases. In phase-1, a wheat barley composite flour shall be developed. Four preparations of the flour shall be developed consisting of pure full grain wheat flour, and three combinations of wheat and barley (W:B) in the ratio of 70:30, 65:35 and 60:40 shall be prepared. Food grade xanthan gum shall be added; 0.5 grams each to all the three wheat barley composites in order to compensate for the gluten loss. All the four flours shall be tested for sensory qualities, rheology, glycemic index, and beta glucan content, and an acceptable composite flour with best attributes shall be further evaluated through proximate analysis. This chosen composite shall be tested in phase-2, in a randomized open label randomized controlled clinical trial in real patients at Akhuwat Medical Center which is a charity facility. The sample size for a power of 90 has been calculated to be 31 and adding for dropouts, rounded up to 35 for each group. 70 Adult non pregnant Type 2 Diabetics above the age of 25, with no serious comorbidity shall be recruited and randomized through computer generated random number table. One group shall receive the 2 kg of composite flour every week for 3 months in addition to usual treatment while the control group shall receive only the usual treatment.

Data collection: BMI, HbA1C, Creatinine, fasting lipid profile and ALT shall be measured at the start and end of the study, while, Fasting and post meal sugars, blood pressure, appetite, satiety, and compliance shall be measured every week. Change in HbA1C from baseline to end of study will be our primary outcome while changes all the other parameters will be our secondary outcomes.

Statistical analysis: The data shall be processed in SPSS 23. HbA1C, BMI, Lipid profile, creatinine and ALT shall be for analysis of Variance (ANOVA), and weakly changes in Fasting and post meal sugars, blood pressure, appetite, satiety and compliance shall be evaluated through factorial analysis to assess the effect of composite flour over time. Both analyses shall be conducted with a Significance Level at P - value < 0.05 for all the parameters Expected outcomes: This study is expected to show a significant improvement in glycemic control with a possible benefit in BP, satiety, weight and lipid profile.

STATEMENT OF THE PROBLEM

Diabetes is a very common chronic disorder across the globe including Pakistan. Poor control of this disease can lead to serious and fatal acute as well as chronic complications. Management of diabetes is however difficult and cumbersome, especially in the sense that it involves continued lifestyle modifications, including dietary constraints and restraints. It would be ideal for people with diabetes to have one such food in their diet, which can manage their diabetes and relieves them of all the bother to manage their every single meal for maintaining a reasonable glycemic control.

This ideal though seems very far at this moment, functional foods and nutraceuticals are a fair step in this direction. Barley due to its high content of the soluble fiber beta glucan has been shown to help glycemic control, but barley does not make good dough, while isolated beta glucan is very expensive to be used in every day diet of the common man.

The Present study is designed with the objective of formulating a nutritionally efficient wheat barley composite flour, which is not only palatable and economical but can replace the wheat flour chapattis in the diet of people with t ype-2 diabetes and will improve their glycemic control simply by this substitution. This effect shall be substantiated through a randomized controlled clinical trial

HYPOTHESIS

Wheat-barley composite flour replaced with wheat in the diet of diabetics will improve their glycemic control

MATERIALS AND METHODS This Study will be conducted in two phases

1. Product development and Nutrient Profiling,
2. Open Label Randomized controlled Clinical Trial in Human Volunteers

PHASE-1 (PRODUCT DEVELOPMENT AND NUTRIENT PROFILING)

Procurement of raw Material

1. Whole grain wheat flour shall be procured from "Rehmat Flour Mills, Ravi Road Lahore
2. Barley Flour Shall be procured from the local grain market, Akbari Mandi Lahore.
3. Food Grade Xanthan Gum shall be Obtained from the local Chemical Market, Shah Aalam Market Lahore.

Product Development Three formulations of the composite flour and one of the whole wheat flour shall be prepared for comparative sensory testing as follows Name Wheat % Barley % Xanthan Gum % A 100 0 0 B 69.5 30 0.05 C 64.5 35 0.05 D 59.5 40 0.05

Sensory Testing Chapattis (flat bread from unleavened flour) shall be made from all the four types of flour, and shall be presented before an expert panel with five numbers, who shall vote for the following characteristics on an interval scale of 1-5 (Basic Sensory Methods for Food Evaluation)

1. Color
2. Odor
3. Texture
4. Taste
5. Overall acceptability

   Rheology Studies Rheology studies shall be conducted for all the four formulations with the help of Rheometer at Rehmat Flour Mills laboratory.

   Glycemic Index Glycemic Index of all the four formulations shall be conducted according to standard international method as described by the Glycemic index foundation (Brouns F et al.,2005).

   The formulation of the flour to be used for the clinical trial shall be selected on the basis of the best match for sensory attributes, the Rheological properties and the glycemic Index. This Chosen formulation shall hitherto be named as "Diaflour"

   Proximate Analysis The Composite flour mixture will be analyzed for moisture, ash, crude protein, crude fiber, crude fat and Nitrogen free extract (NFC) according to their respective methods (AOAC, 2019) Mineral Contents Minerals Like Na, Ca, and K will be estimated by flame photometer according to the procedures of AOAC (2006).

   Beta-Glucan Content The Beta-glucan content of the selected Diaflour shall also be determined through standard methods PHASE-2 (OPEN LABEL RANDOMIZED CONTROL CLINICAL TRIAL)

   An open label randomized controlled clinical trial shall be conducted on real patients of type-2 Diabetes patients at the Diabetic Clinic of Akhuwat Medical Center Township Lahore which is a charity Diabetes service Sample size calculation Sample size has been calculated according to Chan's method (Chan, 2003). We used Table |II of Page 174 with the parameter delta =0.9 with 90% power of the test for rejecting the false hypothesis, which requires 27 participants in both groups. Adding up for drop-outs, we have rounded up the figure 35+35 Participants Seventy consecutive consenting volunteers shall be recruited over a period of 3 months according to the following criteria A. Inclusion Criteria
   1. People with Type-2 Diabetes of any duration
   2. Age ≥ 25
   3. Consenting to participate B. Exclusion Criteria

   <!-- -->

   1. People with Type-1 Diabetes
   2. All pregnant Ladies
   3. Any serious comorbidity unrelated to diabetes on clinical evaluation
   4. People with advanced kidney and liver disease Randomization The enrolled participants shall be randomized according to computer generated random numbers table and divided in to two groups A. Diaflour Group B. Usual Treatment Group Treatment A. Composite Flour Group The composite flour (treatment) group shall continue to receive the usual treatment suggested by their physician along with any changes that the physician deems necessary during the 3 month period of this study. They will additionally receive 2 Kg of the composite flour every week, sufficient for 21 chapattis, and shall eat chapattis made from this flour instead of their usual wheat flour chapattis.

   B. Usual Treatment Group This group shall receive only the usual treatment suggested by their physician along with any changes that the physician deems necessary during the 3 month period of this study. They will continue to eat their usual diet as before their enrollment. They shall however receive usual counseling on lifestyle modifications including diet.

   Data Collection The Following data shall be collected during the study Parameter Time Height Baseline only Weight & BMI Baseline and end of study Appetite Weekly Satiety Weekly Compliance with provided treatment Weekly BP Weekly Fasting Blood Sugar Weekly Post Meal Sugar Weekly HbA1C Baseline and end of study Fasting Lipid Profile Baseline and end of study Creatinine Baseline and end of study ALT Baseline and end of study Parameter Time

   Duration of the Study This project shall be completed in a period of 15 to 18 months, and the time taken for each segment is expected to go as follows Phase -1 3 months Phase-2 Enrollment 3 months Run-in (Washout) Period 2 weeks Treatment period 3 months Lab work and data analysis 3 months Write -up 3 months Total Duration 15.5 months

   Data Analysis Statistical analysis: The data shall be processed in SPSS 23. HbA1C, BMI, Lipid profile, creatinine and ALT shall be for analysis of Variance (ANOVA), and weakly changes in Fasting and post meal sugars, blood pressure, appetite, satiety and compliance shall be evaluated through factorial analysis to assess the effect of composite flour over time. Both analyses shall be conducted with a Significance Level at P - value < 0.05 for all the parameters Expected outcomes: This study is expected to show a significant improvement in glycemic control with a possible benefit in BP, satiety, weight and

ELIGIBILITY:
Inclusion Criteria:

1. People with Type-2 Diabetes of any duration
2. Age ≥ 25
3. Consenting to participate

Exclusion Criteria:

1. People with Type-1 Diabetes
2. All pregnant Ladies
3. Any serious comorbidity unrelated to diabetes on clinical evaluation
4. People with advanced kidney and liver disease

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in Glycated hemoglobin (HbA1C) | 3 months
  Glycated hemoglobin shall be measured at the time of enrollment and at the end of 3 month of intervention period
Reduction in mean fasting blood sugar | Weekly for three months
  Fasting blood sugar shall be measured every weak
Reduction in 2 hours post meal blood sugar | Weekly for three months
  2 hours post meal sugar shall be measured every week

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asif Mahmood, MCPS, Principal Investigator — Student at University of Veterinary and Animal Sciences
Locations (1):
- Akhuwat Medical Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No